CLINICAL TRIAL: NCT00358202
Title: Phase 4 Study of Once-Daily Intramuscular Cefepime Versus Ceftriaxone for In-Home Treatment of Nursing Home-Acquired Pneumonia
Brief Title: Cefepime vs. Ceftriaxone to Treat Nursing Home-Acquired Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CPL Associates (Other)
Collaborators: Elan Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NUR0300202A
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Pneumonia
Keywords: intramuscular antibiotics; nursing home acquired pneumonia; nhap; pharmacoeconomics; cefepime; ceftriaxone
MeSH Terms: conditions — Pneumonia | interventions — Cefepime; Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 cefepime (Active Comparator)
  Interventions: Drug: cefepime
- 2 ceftriaxone (Active Comparator)
  Interventions: Drug: ceftriaxone

INTERVENTIONS:
Drug: cefepime — cefepime hydrochloride 1gm IM q24h
  Arms: 1 cefepime
Drug: ceftriaxone — ceftriaxone 1 gm IM q24h
  Arms: 2 ceftriaxone

SUMMARY:
Randomized trial of nursing home residents with pneumonia to assess if intramuscular cefepime is a safe, efficacious, and cost-effective alternative to once daily intramuscular ceftriaxone for the treatment of elderly nursing home residents who develop pneumonia and do not require hospitalization.

DETAILED DESCRIPTION:
To compare the efficacy, safety, and pharmacoeconomics of cefepime versus ceftriaxone. Double-blind study of nursing home residents >60 years of age with pneumonia. Patients were randomized to cefepime or ceftriaxone 1 gm q24h to be administered intramuscularly. After three days, responding patients could be switched to oral antibiotics. Main Outcome Measures: clinical success, adverse events, and cost-effectiveness ratios.

ELIGIBILITY:
Inclusion Criteria: Residents of a nursing home for >=30 days who were at least 60 years of age and developed pneumonia not amenable to oral antibiotics while not requiring hospitalization, a new infiltrate on chest Xray, estimated Clcr <=60 mL/min, presence of standard clinical criteria, signed informed consent.

Exclusion Criteria: Allergy to cephalosporins, receipt of >24 hours of an antibiotic (unless no improvement was evident), an existing infection due to a pathogen known resistant to either study drug; expected mortality within 48 hours, immunosuppression, hypotension or respiratory distress requiring ventilatory support, prior limited treatment or supportive care only directives, suspected or known Pseudomonas aeruginosa or MRSA infections, primary lung cancer or another malignancy metastatic to the lungs, bronchial obstruction or a history of post-obstructive pneumonia, or patients receiving renal dialysis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2002-03; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Total cost of all antibiotics. | 7-14 days

SECONDARY OUTCOMES:
Clinical efficacy, safety, and cost-effectiveness analysis of total healthcare costs. | 7-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Paladino, PharmD, Principal Investigator — CPL Associates, LLC
Locations (1):
- CPL Associates,LLC, Buffalo, New York, United States